CLINICAL TRIAL: NCT04365374
Title: A Phase 3 Randomized Controlled Trial of Post-Surgical Stereotactic Radiotherapy (SRT) Versus Surgically Targeted Radiation Therapy (STaRT) With Gamma Tile for Treatment of Newly Diagnosed Metastatic Brain Tumors.
Brief Title: Post-Surgical Stereotactic Radiotherapy (SRT) Versus GammaTile-ROADS (Radiation One and Done Study)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GT Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTM-102
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Brain Metastases
Keywords: Brain; Tumor; Cancer; New Diagnosis; Metastases; GammaTile; Radiation; Cs-131
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgical Resection and GammaTile Therapy (Experimental): Surgical Resection and GammaTile Therapy
  Interventions: Device: Gamma Tile-Surgically Targeted Radiation Therapy (STaRT)
- Surgical Resection and Stereotactic Radiation Therapy (Active Comparator): Surgical Resection and Stereotactic Radiation Therapy
  Interventions: Radiation: Stereotactic Radiation Therapy

INTERVENTIONS:
Device: Gamma Tile-Surgically Targeted Radiation Therapy (STaRT) — GammaTiles are a permanently implanted radiation device consisting of Cs-131 seeds positioned within a collagen tile
  Other Names: Carrier Tile Brachytherapy Therapy (CTBT)
  Arms: Surgical Resection and GammaTile Therapy
Radiation: Stereotactic Radiation Therapy — External Beam Radiation Therapy
  Arms: Surgical Resection and Stereotactic Radiation Therapy

SUMMARY:
This trial will be a randomized controlled study comparing the efficacy and safety of intraoperative radiation therapy using GammaTilesTM (GT) versus SRT 3-4 weeks following metastatic tumor resection which is the current standard of care.

DETAILED DESCRIPTION:
GammaTile therapy results in improved clinical outcomes; however, the data is a single site experience with a limited number of subjects, including only 12 of which were patients with metastatic brain tumors. The primary objective of this randomized, controlled trial is to compare the efficacy and safety of intraoperative radiation therapy using GammaTile® (GT) versus SRT 3-4 weeks following metastatic tumor resection which is the current standard of care. The data collected in this trial design will allow for a direct comparison of a variety of outcomes including local control, overall survival, functional status, quality of life, neurocognitive status, and safety in the target population. In order to support direct comparisons, subjects will be randomized to the two equally sized arms (1:1) based on the following stratification factors: age (<60 vs ≥60), duration of extracranial disease control (≤3 months vs >3 months), number of metastases (one, 2-4 total, 5-6 total ), histology (breast cancer, lung cancer, melanoma, other), the maximal diameter of the index lesion (≤3 cm, >3 cm to ≤5cm, >5cm to ≤7cm) and use of prior or current immunotherapy (yes vs no).

An index lesion meeting the criteria of ≥ 2.0-7.0 cm in maximum diameter and appropriate for gross total resection (GTR), will be identified and up to five (5) other unresected, previously untreated lesions in a patient will be allowed. After resection of the index lesion, the surgical bed will be treated with adjunct radiation (either GT or SRT) thereby following the standard of care guidelines (NCCN Guidelines, 2019). Additionally, all unresected, previously untreated metastatic lesions will be treated with stereotactic radiosurgery alone, which also adheres to standard of care guidelines (NCCN Guidelines, 2019).

GammaTile is an FDA-cleared means of rapid dose delivery of radiation therapy directly to the tumor bed with predictable dosimetry at the immediate time of resection, and an intense but localized radiation treatment may confer a reduced risk for radiation necrosis compared to other therapies. It is typically easily placed with minimal additional operative time and limited staff radiation exposure.

Given these benefits, the rationale for conducting this randomized controlled comparison study is to generate additional data, to further support the use of this new FDA-cleared method of delivering radiation therapy in the setting of newly diagnosed brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years old and above. Eligibility is restricted to this age group given that the battery of neurocognitive tests utilized in this protocol are not developed or validated for use in a younger population.
2. One to six newly diagnosed brain metastases, identified on the screening MRI, from an extracranial primary tumor.
3. Only one lesion, designated the index lesion, is planned for surgical resection. The index lesion must be between 2.0 and 7.0 cm in maximal extent on the screening MRI, and gross total resection is expected by the neurosurgeon.
4. Non-index lesions must measure ≤ 4.0 cm in maximal extent on the screening MRI brain scan. The unresected lesions will be treated with SRT as outlined in the treatment section of the concept.
5. All metastases must be located ≥ 5 mm from the optic chiasm and outside the brainstem. Dural based metastasis are eligible.
6. Previous and/or concurrent treatment with investigational or FDA approved systemic therapies (e.g., chemotherapy, targeted therapeutics, immunotherapy) are permitted and must follow protocol guidelines as follows: Systemic therapy is allowed a minimum of one week from last systemic therapy cycle to surgical resection, and one week after surgical resection to allow a minimum of one week before starting/resuming systemic therapy, depending on the specific systemic agent(s), as recommended by medical/neuro-oncology. Systemic therapy is not allowed 1 day before SRT, the same day as the SRT, or 1 day after the completion of the SRT or longer, depending on the specific systemic agent(s), as recommended by medical/neuro-oncology. Agents that are delivered by implant or depot injections (such as hormonal therapies) are excluded from these restrictions.
7. Karnofsky Performance Scale (KPS) score of ≥ 70. Patients with KPS < 70 can be enrolled if their baseline KPS within 14 days of screening was estimated ≥ 70 and surgical management is expected to improve KPS to ≥ 70.
8. Stable systemic disease or reasonable systemic treatment options predicting a life expectancy of ≥6 months.
9. Ability to complete an MRI of the head with contrast
10. Adequate renal and hepatic function to undergo surgery, in investigators opinion.
11. For women of childbearing potential only, a negative urine or serum pregnancy test done <7 days prior to randomization is required. Women must be willing to notify investigator immediately if they become pregnant at any time during the trial period.
12. Men and women of childbearing potential must be willing to employ adequate contraception throughout the study and for men for up to 3 months after completing treatment.
13. Subjects must be fluent in English, Spanish, or another language the study site is prepared to obtain informed consent for in this trial. English speaking subjects will complete Neurocognitive assessments. Non-English-speaking subjects are trial-eligible but will not complete the Neurocognitive assessments as the psychometric properties for translated tests are either not known or not as robust.
14. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedures. A legally authorized representative may provide consent if the potential subject lacks the capacity to provide consent themselves.

Exclusion Criteria

1. Age <18 years.
2. Karnofsky Performance Scale (KPS) score of <70. Patients with KPS < 70 can be enrolled if their baseline KPS within 14 days of screening was estimated ≥ 70 and surgical management is expected to improve KPS to ≥ 70.
3. Sensitivity to bovine (cow) derived materials including collagen products.
4. Past radiation or surgical therapy to the index lesion or the newly diagnosed non-index lesion(s) is exclusionary. However, up to a total of 2 prior courses of SRT treatment to previously diagnosed lesions are allowed as long as any treated lesions are were ≥15mm from the index lesion.
5. Patients with >6 newly diagnosed metastases on screening MRI
6. Pregnant patients.
7. Primary germ cell tumor, small cell carcinoma, or lymphoma.
8. Leptomeningeal metastasis (LMD). Note: For the purposes of exclusion, LMD is a clinical diagnosis, defined as radiologic or clinical evidence of leptomeningeal involvement with or without positive cerebrospinal fluid (CSF) cytology.
9. Prior WBRT for brain metastases.
10. Concomitant therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
11. Comorbid psychiatric or neurologic disease or injury impacting cognition, in the opinion of the treating physician, that might impair patient's ability to understand or comply with the requirements of the study or to provide consent
12. Subjects who, in the investigator's opinion, are unable to understand the protocol or to give informed consent, have a history of poor cooperation, noncompliance with medical treatment, or difficulty in returning for follow up care. A legally authorized representative may provide consent if the potential subject lacks the capacity to provide consent themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Surgical bed recurrence-free survival (SB-RFS) from the time of randomization up to 2 years post radiation. | up to 2 years post-radiation
  Surgical bed control is defined as the absence of new nodular contrast enhancement in the index lesion surgical bed.

SECONDARY OUTCOMES:
Overall Survival | up to 3 years
  Survival of subjects
Functional Assessment of Cancer Therapy-Brain (FACT-Br) | up to 9 months
  An assessment of quality of life (QOL)
Linear Analog Scale Assessments (LASA) | up to 9 months
  An assessment of quality of life (QOL)
Hopkins Verbal Learning Test (HVLT-R) | up to 24 months
  An assessment of neurocognitive status
Controlled Oral Word Association Test (COWAT) | up to 24 months
  An assessment of neurocognitive status
Trail Making Tests (TMT) Parts A and B | up to 24 months
  An assessment of neurocognitive status
Barthel ADL | up to 24 months
  An assessment of physical functioning status

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weinberg, MD, Principal Investigator — MD Anderson Cancer Center, Houston, TX
Locations (37):
- United States (37):
  - HonorHeath Scottsdale Osborn Medical Center, Phoenix, Arizona
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - Ascension St. Vincent's- Riverside, Jacksonville, Florida
  - Baptist MD Anderson Cancer Center- Jacksonville, Jacksonville, Florida
  - HCA Florida First Coast Neurology- Orange Park, Orange Park, Florida
  - Advent health Orlando, Orlando, Florida
  - Orlando Health, Orlando, Florida
  - Florida Health Sciences Center, Inc. d/b/a Tampa General Hospital, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - RUSH University, Chicago, Illinois
  - Indiana University, IU Health Methodist Hospital, Indianapolis, Indiana
  - The University Of Kansas Cancer Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri, Columbia, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - HMH Jersey Shore University Medical Center, Neptune City, New Jersey
  - Albany Medical Center, Albany, New York
  - Memorial Sloan Kettering, New York, New York
  - Westchester Medical Center, Westchester, New York
  - University of North Carolina Health, Chapel Hill, North Carolina
  - ECU Health, Greenville, North Carolina
  - Mayfield Brain and Spine, Cincinnati, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Brown University Health, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Simmons Cancer Center, Dallas, Texas
  - Baylor St. Luke's Medical Center | Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - SCRI with Texas Oncology, The Woodlands, Texas
  - Virginia Mason, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weinberg J. Clinical Trials in Progress: ROADS Trial. Oncology (Williston Park). 2021 Aug 8;35(8):495. doi: 10.46883/ONC.2021.3508.0495. PMID 34398588